CLINICAL TRIAL: NCT03833310
Title: Novel Biomarkers in Diagnosis of Inflammatory Bowel Disease
Brief Title: Novel Biomarkers in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nesma Gamal, principal investigator, Assiut University
Other Study IDs: vosrd
Record Dates: First submitted 2019-01-14; First posted 2019-02-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2020-05

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — serum specimen from patient with inflammatory bowel disease after diagnosis and healthy persons .second sample taking 3month after received treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Osteoprotegerin, sRANKL, NfKB and TFF3 markers in serum in inflammatory bowel disease — I will measure Osteoprotegerin , Soluble Receptor activator of nuclear factor kappa-Β ligand, Nuclear factor kappa-light-chain-enhancer of activated B cells and Trefoil factor 3 in serum of patient with inflammatory bowel disease

SUMMARY:
The inflammatory bowel diseases represent a heterogeneous group of chronic , relapsing- inflammatory disorders of the gastrointestinal tract. Crohn's disease and ulcerative colitis are the two major clinical forms. Considerable effort has been devoted to the development of an accurate ,noninvasive biomarkers that have increased diagnostic sensitivity and specificity .

Osteoprotegerin is a member of the Tumor Necrosis Factor Receptor superfamily of proteins. I is of particular importance in bone metabolism, inflammation , tumorigenesis, and other processes where cell differentiation, survival, and death are controlled.

Soluble Receptor activator of nuclear factor kappa-Β ligand is known as a type II membrane protein and as a member of tumor necrosis factor superfamily . Soluble Receptor activator of nuclear factor kappa-Β ligand has been identified to affect the immune system and a binding partner of ( Osteoprotegerin ), and controls cell proliferation.

NF-κB is a transcription factor that activates inhibitor of kappa B kinase in the cytosol upon being stimulated by inflammatory stimuli with subsequent signaling pathways via canonical or non-canonical lead to migration of NF-κB toward the nucleus and hence initiates the targeting gene such as pro-inflammatory cells.

TFF3 is predominantly expressed in the goblet cells of the small intestine and colon . Trefoil factor 3 has a key role in mucosal defense and restitution in the gastrointestinal mucosa. It has an anti-apoptotic effect on intestinal epithelial cells. Moreover, it contributes to the stabilization and maintenance of the intestinal epithelial barrier function by simulating the recovery of tight junction proteins .

DETAILED DESCRIPTION:
The inflammatory bowel diseases represent a heterogeneous group of chronic , relapsing-remitting inflammatory disorders of the gastrointestinal tract, and Crohn's disease and ulcerative colitis are among the two major clinical forms The global incidence and prevalence of The inflammatory bowel diseases has increased over the last 2-4 decades, likely because of the adoption of a more "western" lifestyle as well as improved detection and awareness . Despite the great progress in understanding the pathogenesis of these diseases, their etiology remains unclear. Genetic, immune, and environmental factors are thought to play a key role .

In the case of Crohn's disease , chronic inﬂammation can be localized in every gastrointestinal tract segment and involves the full thickness of the intestinal wall. In contrast ,in ulcerative colitis , mucosa and submucosa membranes of the large intestine are usually involved The illness starts in the rectum and generally extends proximally through the whole colon. . Both diseases differ in the localization and size of the segment involved. There are also differences in clinical image, laboratory test results, and different characteristics of complications. The course and grade of disease activity depend on many factors, such as environmental influences , genetic features, changes in the intestinal microbiota ecosystem, and immune factors .

The correct diagnosis of non-specific inflammatory bowel diseases as well as the determination of disease activity, risk stratification , and prediction of response to therapy still relies on a multidisciplinary approach based on clinical, laboratory, endoscopic, and histologic examination . However, considerable effort has been devoted to the development of an accurate panel of noninvasive bio markers that have increased diagnostic sensitivity and specificity .

Osteoprotegerin , also known as is a member of the Tumor Necrosis Factor Receptor superfamily of proteins. Osteoprotegerin is involved in many biological processes: its role is of particular importance in bone metabolism, inflammation , tumorigenesis, and other processes where cell differentiation, survival, and death are controlled. Osteoprotegerin was detected in serum, mucosal biopsies, and in the stool .

The Osteoprotegerin gene is located on chromosome 8q23- 24.17. The mature OPG protein contains 380 amino acids and consists of seven domains. The ﬁrst four domains (D1-D4) contain cysteine-rich structures at the N terminus which are required for the inhibition of osteoclast differentiation. The ﬁfth and the sixth domain (D5 and D6) are death-domains and may be important in cytotoxic signals. The seventh domain, a C terminus heparin-binding site, is involved in dimer osteoprotegerin formation .

Osteoprotegerin can be produced by a wide range of cell types, including osteoblasts, B lymphocytes, dendritic cells, bone marrow stromal cells, epithelial cells, and monocytes/macrophages. Osteoprotegerin activates and/or perpetuates inflammation in the gut by stimulating immune cells, cytokines, and the Necrosis factor-kappa B pathway .

On the other hand, soluble Receptor activator of nuclear factor kappa-Β ligand , also known as tumor necrosis factor ligand. soluble Receptor activator of nuclear factor kappa-Β ligand is known as a type II membrane protein and as a member of tumor necrosis factor superfamily.

Soluble Receptor activator of nuclear factor kappa-Β ligand has been identified to affect the immune system and control bone regeneration and remodeling, a binding partner of , and controls cell proliferation. it is expressed in several tissues and organs including: skeletal muscle, thymus, liver, colon, small intestine, adrenal gland, osteoblast, mammary gland epithelial cells, prostate and pancreas. Variation in concentration levels of soluble Receptor activator of nuclear factor kappa-Β ligand throughout several organs reconfirms the importance of in tissue soluble Receptor activator of nuclear factor kappa-Β ligand growth (particularly bone growth) and immune functions within the body .

The interactions between ,Osteoprotegerin,soluble Receptor activator of nuclear factor kappa-Β ligand and soluble Receptor activator of nuclear factor kappa-Β also have relevance to inflammatory pathways. - soluble binding Receptor activator of nuclear factor kappa-Β binding activates several pathways that contribute to the survival of T-lymphocytes and dendritic cells .

In addition, Osteoprotegerin is synthesized by dendritic and B-lymphocytes whereas soluble Receptor activator of nuclear factor kappa-Β ligand is mainly produced by T-lymphocytes. Moreover, soluble Receptor activator of nuclear factor kappa-Β ligand and various cytokines e.g. Tumor Necrosis Factor α induce the synthesis of osteoprotegerin from immune cells. In turn, the interruption of soluble Receptor activator of nuclear factor kappa-Β - soluble Receptor activator of nuclear factor kappa-Β ligand ligation by osteoprotegerin down regulates T-lymphocyte and dendritic activity, thereby modulating inﬂammatory responses .

Soluble receptor activator of nuclear factor-κB ligand (NF-κB) is a transcription factor that activates inhibitor of kappa B (IκB) kinase in the cytosol upon being stimulated by inflammatory stimuli with subsequent signaling pathways via canonical or non-canonical lead to migration of NF-κB toward the nucleus and hence initiates the targeting gene such as pro-inflammatory cells, monocytes, macrophages, T and B cells (7).

Trefoil factors (TFFFs) comprise a unique family of abundant gastrointestinal peptides with a distinct three-loop structure formed by a highly conserved motif of cysteine disulfide bonds. They are extremely stable against proteolytic digestion and acid degradation. The trefoil factor family consists of three members: TFF1 (breast cancer-associated peptide), TFF2 (spasmolytic polypeptide) and TFF3 (intestinal trefoil factor). TFF3 is predominantly expressed in the goblet cells of the small intestine and colon (8). Trefoil factor 3 has a key role in mucosal defense and restitution in the gastrointestinal mucosa. It has an anti-apoptotic effect on intestinal epithelial cells. Moreover, it contributes to the stabilization and maintenance of the intestinal epithelial barrier function by simulating the recovery of tight junction proteins (9).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients (untreated) by clinical and endoscopic examination and not received treatment .

Exclusion Criteria:

* patients have autoimmune diseases
* patients with cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: After standardized work-up with clinical, endoscopic, histopathologicial and, when applicable, radiological evaluation, all patients will met the generally accepted international diagnostic criteria of inflamatory bowel diseaes .The healthy controls consisted of an age- and gender-matched (negative for IBD). This group did not show evidence or familial history of IBD or any other immune mediated disorders
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
level of Osteoprotegerin, sRANKL, NF kappaB and TFF3 in newly diagnosed patients with inflammatory bowel disease | 2 years
  measuring level of Osteoprotegerin , sRANKL, NFkappaB and TFF3 in newly diagnosed patients with inflammatory bowel disease then it will measured again after treated with corticosteroid and immune therapy or inflximab and immune therapy

CONTACTS AND LOCATIONS:
Overall Officials: nesma gamal, demonstrator, Principal Investigator — Assiut University; ragaa salama, professor, Study Director — Assiut University; Amira Abdel Hamid Kamal Mohamed, Lecture, Study Director — Assiut University; Mohammed Ahmed Medhat, Lecture, Study Director — Assiut University
Locations (1):
- Assuit Medical University, Asyut, Egypt